CLINICAL TRIAL: NCT07271498
Title: "Oral Chronic Graft-Versus-Host Disease (cGVHD) as a Potential Clinical Marker of the Graft-Versus-Leukemia (GVL) Effect in Allogeneic Hematopoietic Stem Cell Transplantation:Prospective Single-Center Study"
Brief Title: The Oral cGVHD as a Predictive Factor of Graft Versus Leukaemia Effect in Patients Who Received an Allograft
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 25Hemato01
Record Dates: First submitted 2025-11-25; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Allografts; Oral cGVHD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with oral cGVHD
  Interventions: Other: Evaluation of oral cGVHD

INTERVENTIONS:
Other: Evaluation of oral cGVHD — analysis statistics

SUMMARY:
Allogeneic hematopoietic stem cell transplantation (allo-HSCT) is the standard treatment for many malignant blood disorders. Its effectiveness is based on the graft-versus-leukemia (GVL) effect, which is intrinsically linked to the occurrence of graft-versus-host disease (GVHD). While GVHD reflects favorable alloreactivity, its severe forms increase While GVHD reflects favorable allograft reactivity, its severe forms increase non-relapse mortality (NRM) and impair quality of life. Currently, there is no simple clinical marker that can predict or monitor the efficacy of the GVL effect. The investigators therefore hypothesized that chronic oral GVHD, a common and easily identifiable manifestation, could reflect beneficial alloreactivity, reflecting a balance between GVL effect and toxicity. The investigators conducted a prospective, observational, single-center study including patients transplanted at the Nice University Hospital between October 2023 and May 2025, followed by a standardized stomatological protocol before and after transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received an allograft between octobre 2023 and May 2025 at CHU de Nice.

Exclusion Criteria:

* Patients who did not received an allograft

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who received an allograft between octobre 2023 and May 2025 at CHU de Nice.
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | 3 months, 6 months, 1 years and 1,5 years
  Overall Survival (OS) is defined as the time, measured in months, from the date of study entry (or randomization, depending on protocol specifications) to death from any cause. Participants who are alive at the time of the last known follow-up are censored at that date.

SECONDARY OUTCOMES:
Disease free survival, | 3 months, 6 months, 1 years and 1,5 years
  Disease-Free Survival (DFS) is defined as the time, measured in months, from the date of curative-intent treatment (or randomization, according to protocol specifications) to the first documented recurrence of the disease or death from any cause, whichever occurs first. Participants who remain alive and free of disease at the time of the last known follow-up are censored at that date.
Non relapse mortality | 3 months, 6 months, 1 years and 1,5 years
  Non-Relapse Mortality (NRM) is defined as the time, measured in months, from the date of allogeneic transplantation (or study entry, depending on protocol specifications) to death without prior disease relapse or progression. Deaths occurring after documented relapse/progression are not counted as NRM events. Participants who are alive without relapse at last follow-up are censored at that date.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de NICE, Nice, Alpes Maritimes, France